CLINICAL TRIAL: NCT04646460
Title: Context Interventions: Social Modeling and Initial Treatment Experience
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 230137
Record Dates: First submitted 2020-11-13; First posted 2020-11-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Placebo Effect; Pain
Keywords: Placebo effect; Social modeling; Conditioning; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Observed Success - Experienced Success (Experimental): This participant group (N=30) will witness a successful placebo during the "observation phase" (i.e. the demonstrator will display reduced pain expressions after receiving the cream) and experience a successful placebo during the "experience phase" (i.e. the experimenter will reduce the intensity of the pain stimuli after applying the cream).
  Interventions: Behavioral: Observed Success; Behavioral: Experienced Success
- Observed Failure - Experienced Failure (Experimental): This participant group (N=30) will witness a failed placebo during the "observation phase" (i.e. the demonstrator will not display reduced pain expressions after receiving the cream) and experience a failed placebo during the "experience phase" (i.e. the experimenter will not reduce the intensity of the pain stimuli after applying the cream).
  Interventions: Behavioral: Observed Failure; Behavioral: Experienced Failure
- Observed Success - Experienced Failure (Experimental): This participant group (N=30) will witness a successful placebo during the "observation phase" (i.e. the demonstrator will not display reduced pain expressions after receiving the cream) and experience a failed placebo during the "experience phase" (i.e. the experimenter will not reduce the intensity of the pain stimuli after applying the cream).
  Interventions: Behavioral: Observed Success; Behavioral: Experienced Failure
- Observed Failure - Experienced Success (Experimental): This participant group (N=30) will witness a successful placebo during the "observation phase" (i.e. the demonstrator will display reduced pain expressions after receiving the cream) and experience a successful placebo during the "experience phase" (i.e. the experimenter will reduce the intensity of the pain stimuli after applying the cream).
  Interventions: Behavioral: Observed Failure; Behavioral: Experienced Success

INTERVENTIONS:
Behavioral: Observed Success — The demonstrator in video gets a placebo treatment, "Levoderm" analgesic cream, which will be shown to be effective at relieving pain.
  Arms: Observed Success - Experienced Failure; Observed Success - Experienced Success
Behavioral: Observed Failure — The demonstrator in the video gets the same placebo treatment, but shows little to no effectiveness from the placebo for relieving pain.
  Arms: Observed Failure - Experienced Failure; Observed Failure - Experienced Success
Behavioral: Experienced Success — The participant will receive reduced stimulus intensities after the placebo cream treatment to reinforce the effectiveness of the cream.
  Arms: Observed Failure - Experienced Success; Observed Success - Experienced Success
Behavioral: Experienced Failure — The participant will not receive reduced stimulus intensities after the placebo treatment, so the cream is not reinforced as effective.
  Arms: Observed Failure - Experienced Failure; Observed Success - Experienced Failure

SUMMARY:
In this experiment, the investigators study the brain pathways underlying several promising context interventions that enhance the strength of placebo effects. Specifically, the investigators examine the separate and joint effects of two of the most powerful context interventions: Social modeling-observing someone else being effectively treated-and prior treatment success or failure experiences. Participants will be randomized into 4 groups (Social modeling: observed success vs. observed failure and Conditioning: experienced success vs. experienced failure). The objectives are to investigate the placebo effect on pain relief and aversive image stimuli between and within-subjects. Each group will undergo a behavioral induction phase, fMRI placebo test phase, and an identical 3-month follow up fMRI placebo test phase. Follow-up assessment will provide some of the first evidence on predictors of the durability of placebo and context interventions.

DETAILED DESCRIPTION:
Background:

Humans are highly social creatures, and others' behavior and experiences can have profound effects on symptoms, physiology, and behavior. Social modeling-watching a similar other experience treatment benefits-may also strongly enhance placebo effects and their durability over time, particularly when combined with other context interventions. Social influences can affect core motivational circuitry (e.g., nAC and amygdala), shape learning trajectories, and appears to have distinct mechanisms from other (e.g., conditioning) manipulations. Their impact on brain mechanisms of placebo has not been studied. Likewise, initial perceived treatment success or failure can powerfully shape learning trajectories and placebo analgesia. Initial failure experiences with a treatment type (e.g., pill) may explain some of the treatment failures in studies that (a) attempt to wash out placebo responses with ineffective pills before starting verum drug, or (b) re-randomize non-responders to different pills, as in the STAR*D antidepressant study. But the effects of initial success/failure experiences on the brain mechanisms of placebo effects have not been studied.

Design:

In an initial observation phase, participants will watch a video of another participant ("demonstrator") undergoing the baseline assessment and placebo test procedure. Next, participants will undergo a conditioning phase. The intervention is a 2 x 2 factorial between-groups manipulation (N = 30 per group) of social modeling (Observed treatment success vs. failure) and participants' initial success experience (Experienced success vs. failure). Thus, the demonstrator will either show strong signs of pain relief during placebo (Observed-Success condition) or no signs of relief (Observed-Failed treatment). During the conditioning phase, all participants will experience high-intensity heat before placebo treatment and then either low-intensity heat after application of a placebo cream, as in the investigator's and others' past work, creating experience of pain relief (Experienced-Success condition) or they will not experience relief (i.e., temperatures will not be lowered; Experienced-Failed treatment). In a subsequent fMRI test phase, participants experience painful heat and aversive IAPS images (as a transfer/specificity test) during fMRI, on skin sites treated with Control and Placebo creams, in a Control -> Placebo -> Control block design as in past research. Finally, a 3-month follow-up fMRI test phase, without additional observation or conditioning, will assess durability of brain and behavioral placebo effects.

ELIGIBILITY:
Inclusion Criteria:

* No current psychiatric or major neurological diagnosis
* No reported substance abuse within the last six months
* Capable of performing experimental tasks (e.g., are able to read, able to cooperate with fMRI examination)
* Fluent or native speakers of English
* No current or recent history of pathological pain or reported neurological disorders
* Abstained from alcohol and substance use for 48 hours
* Provided informed consent
* Passed fMRI screening test

Exclusion Criteria:

* Current presence of pain
* Current or past history of primary psychiatric disorder
* Current or past history of psychoactive substance abuse or dependence
* Dementias
* Movement disorders except familial tremor
* CNS infection
* CNS vasculitis, inflammatory disease or autoimmune disease
* CNS demyelinating disease (e.g. multiple sclerosis)
* Space occupying lesions (mass lesions, tumors)
* Congenital CNS abnormality (e.g. cerebral palsy)
* Seizure disorder
* History of closed head trauma with loss of consciousness
* History of cerebrovascular disease (stroke, TIAs)
* Abnormal MRI (except changes accounted for by technical factors or UBOs)
* Neuroendocrine disorders (e.g., Cushings disease)
* Uncorrected hypothyroidism or hyperthyroidism
* Current or past history of cancer
* Recent history (within two years) of myocardial infarction, severe cardiovascular disease, or currently active cardiovascular disease (e.g. angina, cardiomyopathy)
* Uncontrolled hypertension or hypotension
* Chronic pain syndromes
* Chronic fatigue syndromes
* Subjects unable to tolerate the scanning procedures (e.g., claustrophobia)
* Prior treatment within the last month with any of the following: antidepressants, mood stabilizers, glucocorticoids, opiates
* Prior treatment with any of the following: antipsychotics, isoniazid, centrally active antihypertensive drugs (e.g. clonidine, reserpine)
* Metal in body or prior history working with metal fragments (e.g., as a machinist)
* Pregnancy
* Any other contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body)
* Claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Intervention effects on pain ratings | Immediately after pain stimuli
  Pain ratings will be given on a 0-100 scale. 0 being "no pain at all" and 100 being "most pain imaginable in the context of this study."
Intervention effects on aversive image ratings | Immediately after aversive image stimuli
  Aversive ratings will be given on a 0-100 scale. 0 being "not unpleasant at all" and 100 being "very unpleasant."
Brain: signature responses to pain and aversive images | Immediately after pain/image stimuli
  A priori regions of interest response from the brain (fMRI) patterns to the pain and aversive images.

SECONDARY OUTCOMES:
Skin conductance | Immediately after pain stimuli
  Skin conductance response (SCR) will be recorded during the task.
Heart rate | Immediately after pain stimuli
  Heart rate will be recorded during the task.
Whole-brain maps of intervention effects | Immediately after pain stimuli
  Exploratory brain analysis will include univariate voxel-wise maps comparing participant groups with a threshold of q < 0.05, False Discovery Rate (FDR)-corrected.
CliexaEase App ratings | Daily for: 2 weeks before scan, 2 weeks after last scan. Weekly for 1 year after last session.
  Participants click an "I feel" button to display a list of feelings (i.e., happiness, sadness, pain, fear, stress, etc.), and then can drag a feeling bubble to a bodily location (or to a location indicating "not felt in the body"), and then rate the intensity of the feeling on a visual analog scale. This assessment is open-ended to minimize demand characteristics.
Interpersonal Reactivity Index | Within two weeks before first fMRI scan
  A rating of dispositional empathy with responses answered on a 5-point Likert scale ranging from "does not describe me well" to "describes me very well." Higher scores indicate more empathetic responses.

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators are strongly committed to contributing to open and reproducible science. All MRI and behavioral data will be submitted to the NIMH Data Archive (NDA) according to the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html ) and with OpenFMRI.
  The investigators will ensure that our IRB has approved our Data Sharing Plan. The investigators will use an informed consent document that permits subjects to allow sharing of de-identified (face removed) MRI and fMRI data with open-sharing repositories, including the NDA and OpenFMRI databases. The consent form will stipulate that: "Scientists can use my information, without personal identifiers, for any kind of genetic research."
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to NDA within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to NDA/OpenFMRI when the primary study manuscript is accepted.
Access Criteria: These data would generally be made available to any qualified investigator for neuroimaging studies only including:
  i. Research on any brain phenomenon; ii. Neuroimaging research on non-disease traits (intelligence, behavioral traits); iii. Methods development research.
  The requesting investigator must provide documentation of local IRB approval.
  These data would not be made available to:
  i. Any criminal justice organization, because data may not be used for any criminal justice applications; ii. Any commercial entity, because use of the data is limited to not-for-profit organizations and data may not be used for any commercial purposes.